CLINICAL TRIAL: NCT00821145
Title: Laparoscopic Aortic Resection Versus Open Surgery in Patients With AAA
Brief Title: Laparoscopic Versus Open Abdominal Aortic Aneurysm (AAA) Exclusion
Acronym: LapAorta
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: inability to recruit sufficient number of patients
Sponsor: Augusta Hospital Duesseldorf (Other)
Collaborators: Storz GmbH FRG (Unknown); Tel Aviv University (Other)
Responsible Party: Ralf Kolvenbach, Prof. M.D., Catholic clinics Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LapAorta2008
Record Dates: First submitted 2009-01-08; First posted 2009-01-13 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2009-01

CONDITIONS: Infra and Juxtarenal Abdominal Aortic Aneurysms
Keywords: abdominal aortic aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 50 patients operated using a conventional open surgery to exclude an abdominal aortic aneurysm
  Interventions: Procedure: conventional surgery
- 2 (Experimental): 50 patients operated using a total laparoscopic aortic aneurysm resection
  Interventions: Procedure: laparoscopic AAA resection
- 3 (Active Comparator): 25 patients using a laparoscopic approach for AAA resection with a stapled proximal anastomosis
  Interventions: Procedure: laparoscopic stapler anastomosis

INTERVENTIONS:
Procedure: conventional surgery — AAA patients operated using a conventional incision
  Arms: 1
Procedure: laparoscopic AAA resection — laparoscopic AAA resection
  Arms: 2
Procedure: laparoscopic stapler anastomosis — laparoscopic AAA resection, proximal anastomosis performed with a stapler
  Arms: 3

SUMMARY:
In many countries the gold standard for treating abdominal aortic aneurysms is still open surgery with a long incision. In patients with suitable anatomy alternatively an endovascular approach can be chosen. Since open surgery is more durable in many countries a laparoscopic procedure using " key hole surgery " has gained wider acceptance. The current study wants to prove that laparoscopic aortic aneurysm procedures are less invasive than open surgery with reduced recovery times.

DETAILED DESCRIPTION:
In many countries the gold standard for treating abdominal aortic aneurysms is still open surgery with a long incision. In patients with suitable anatomy alternatively an endovascular approach can be chosen. Since open surgery is more durable in many countries a laparoscopic procedure using " key hole surgery " has gained wider acceptance. The current study wants to prove that laparoscopic aortic aneurysm procedures are less invasive than open surgery with reduced recovery times.

Study design: Multi center prospective randomized study including patients with infra or juxtarenal aortic aneurysms ( AAA).

In group I the AAA is resected using a conventional long incision and standard procedures for resecting the AAA. A Dacron graft is used in inlay technique to restore blood flow.

In group II a total laparoscopic approach is chosen to exclude the AAA. Identical to open surgery a dacron graft is laparoscopically sawn in to exclude the AAA and to restore blood flow.

In a subgroup II a the laparoscopic anastomosis is performed with a stapling device to simplify and to accelerate the procedure.

Endpoints of the study:

Total operating time, aortic crossclamping time, stay in ICU, return to a regular diet,postoperative ileus, total hospital stay, major and minor complications, blood loss, renal function in cases with juxtarenal AAA.Patients are evaluated for postoperative pain, wound related problems, hernias and time until full mobilisation is achieved.

Hypothesis: The laparoscopic approach though associated with a longer operating time and longer clamping times is associated with a reduced recovery time, les pain and less wound related problems compared to a full length conventional incision.

ELIGIBILITY:
Inclusion Criteria:

* patients with abdominal aortic aneurysms
* fit for open surgery

Exclusion Criteria:

* patients unfit for open surgery
* patients with malignancies

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
All cause mortality, reduced recovery postoperatively according to pain measurement, ICU and hospital stay, minor and major complications | 1 year

SECONDARY OUTCOMES:
Use of a stapling device reduces total operative time and crossclamping period | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ralf R Kolvenbach, M.D.PhD, Principal Investigator — Augusta Hospital Duesseldorf